CLINICAL TRIAL: NCT06844448
Title: The Effect of Different Risk Factors on the Success Rate of VPT: an Observational Prospective Cohort Study
Brief Title: The Effect of Different Risk Factors on the Success Rate of VPT
Status: Recruiting | Type: Observational
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Dr. Vag Janos, Professor, Semmelweis University
Other Study IDs: 885
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Dental Caries Extending to Pulp; Pulp Disease, Dental; Irreversible Pulpitis; Reversible Pulpitis; Pulpitis
MeSH Terms: conditions — Dental Pulp Diseases; Pulpitis | interventions — tricalcium silicate; Septodont; Pemetrexed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- direct pulp capping: After local anaesthesia the tooth is absolutely isolated. The coronal part of the tooth is then disinfected with a cotton pellet soaked in 5% sodium hypochlorite. Under an operating microscope, the caries is removed non-selectively towards the pulpal wall. The absence of caries on non-pulpal walls is confirmed by caries indicator. The pulp chamber is opened with a sterile diamond bur in a turbine with copious water cooling. After opening the pulp gentle pressure of a sterile cotton pellet soaked in 2.5% NaOCl is applied to the exposed pulp to achieve hemostasis.
  Interventions: Procedure: with Biodentine; Procedure: with MTA
- partial pulpotomy: After local anaesthesia the tooth is absolutely isolated. The coronal part of the tooth is then disinfected with a cotton pellet soaked in 5% sodium hypochlorite. Under an operating microscope, the caries is removed non-selectively towards the pulpal wall. The absence of caries on non-pulpal walls is confirmed by caries indicator. The pulp chamber is opened with a sterile diamond bur in a turbine with copious water cooling. After opening of the pulp with a sterile diamond bur, an additional 2-3 mm of coronal pulp tissue is removed with copious water cooling. Subsequently, light pressure is applied to the pulp for 5 minutes with a cotton pellet dipped in 2.5% NaOCl to control bleeding.
  Interventions: Procedure: with Biodentine; Procedure: with MTA
- complete pulpotomy: After local anaesthesia the tooth is absolutely isolated. The coronal part of the tooth is then disinfected with a cotton pellet soaked in 5% sodium hypochlorite. Under an operating microscope, the caries is removed non-selectively towards the pulpal wall. The absence of caries on non-pulpal walls is confirmed by caries indicator. After the coronal pulp tissue is removed down to the level of the orifices using a sterile diamond bur with copious water cooling. Bleeding is controlled by gentle pressure with a cotton pellet soaked in 2.5% NaOCl.
  Interventions: Procedure: with Biodentine; Procedure: with MTA

INTERVENTIONS:
Procedure: with Biodentine — After the bleeding has stopped, the cavity is flushed with sterile saline and Biodentine (Septodont, Saint-Maur-des-Fossés, France) is mixed according to the manufacturer's instructions. First it is applied directly to the pulp wound using light pressure, and then the entire cavity is filled with it. One week later the superficial 2-3 mm is removed and replaced it with permanent restoration.
  Other Names: Biodentine, Septodont
Procedure: with MTA — After the bleeding has stopped, the cavity is flushed with sterile saline and MTA+ (Cercamed, Stalowa Wola, Poland) is mixed according to the manufacturer's instructions. First it is applied directly to the pulp wound using light pressure, and after its initial setting the cavity is filled with glass ionomer cement. One week later the glass ionomer cement is removed and replaced it with permanent restoration.
  Other Names: MTA +, Cercamed

SUMMARY:
This study aims to evaluate the effectiveness of various vital pulp therapy (VPT) methods, such as direct pulp capping, partial pulpotomy, and total pulpotomy, in maintaining pulp vitality following pulp exposure. It explores the success rates of these treatments compared and investigates co-factors influencing these rates, including age. This prospective cohort study involves patients over 18 with restorable teeth and exposed pulp chambers. Success is measured through clinical and radiological criteria over a follow-up period of up to four years. The study also aims to identify if there's an age threshold affecting the preference for VPT over root canal therapy.

DETAILED DESCRIPTION:
Objectives: The primary objective of this study is to explore the effectiveness of different VPT methods after pulp exposure. A secondary objective is to establish the relationship between success rate, age and other co-factors.

Study methodology: We plan a single-centre, three-arm, observational prospective cohort study. The study will be organised and hosted by the Department of Restorative Dentistry and Endodontics, Semmelweis University. Patients for the study will be selected from patients presenting at the ambulance of the Semmelweis University Department of Restorative Dentistry and Endodontics.

For patients who meet the inclusion criteria, we record the patient's baseline clinical data Baseline data, as well as information obtained during the study and findings during follow-up (7 days, 6 months, 1 year, 2 years, 3 years, 4 years) are recorded by the interventionalist in an online database (REDCap).

Interventions are carried out according to the following steps: After local anaesthesia (Lidocaine-adrenaline 20 mg/0.01 mg/ml, Egis, Budapest, Hungary) and mouth rinsing with 0.2% chlorhexidine, the tooth is absolutely isolated using a rubber dam and liquid dam (Opaldam- Ultradent, South-Jordan, Utah). The coronal part of the tooth is then disinfected with a cotton pellet soaked in 5% sodium hypochlorite (NaOCl). Under an operating microscope, the caries is removed non-selectively, first with a diamond bur under water cooling, then with a steel bur inserted in a handpiece, moving from the periphery of the tooth towards the pulpal wall. The absence of caries on non-pulpal walls is confirmed by caries indicator (Sable Seek-Ultradent, South-Jordan, Utah). The pulp chamber is opened with a sterile diamond bur in a turbine with copious water cooling. After opening the pulp, different types of treatment are used depending on the extent of inflammation and caries.

1. Direct pulp capping: Pressure of a sterile cotton pellet soaked in 2.5% NaOCl is applied to the exposed pulp to achieve hemostasis. After the bleeding has stopped, the cavity is flushed with sterile saline and Biodentine (Septodont, Saint-Maur-des-Fossés, France) or MTA is mixed according to the manufacturer's instructions. The patient is called back after 1 week, when the temporary restoration is removed and a final restoration is placed in the cavity, which may be a composite filling, inlay or crown, depending on the amount of remaining tooth material. This type of intervention is performed (1) if a healthy tooth with a normal pulp has suffered iatrogenic pulp exposure and the pulp tissue is surrounded by intact dentin tissue, and (2) when it is asymptomatic, or with reversible pulpitis symptoms after extra deep caries removal, there is no dentin chips are the pulp tissue, it is surrounded by healthy dentin, there is no evidence of necrosis in the pulp, and bleeding can be controlled within 5 minutes with a cotton pellet soaked in 2.5% NaOCl. Direct pulp capping will berejected if the patient has spontaneous pain before treatment, bleeding from the pulp is not controllable within 5 minutes, necrotic tissue is present in the pulp chamber, or if the pulp is explose through carious dentin.
2. Partial pulpotomy After opening of the pulp with a sterile diamond bur, an additional 2-3 mm of coronal pulp tissue is removed with copious water cooling. Subsequently, light pressure is applied to the pulp for 5 minutes with a cotton pellet dipped in 2.5% NaOCl to control bleeding. After controlling the bleeding, the cavity is flushed with sterile saline and Biodentine or MTA is applied the same way as in case of direct pulp capping. Partial pulpotomy is the treatment of choice in the following clinical situations: (1) in case of extra-deep caries the bacterial biofilm and infected dentin can be only removed by superficial pulp excision, (2) when further caries removal is required after pulp exposure due to the risk of infected dentin shavings entering the pulp, (3) in the case of normal pulp after extra-deep caries removal, bleeding cannot be controlled within 5 minutes after direct pulp capping attempt, (4) in the case of reversible pulpitis, if bleeding cannot be stopped within 5 minutes after pulp exposure. We exclude from partial pulpotomy treatment, for any of the above indications, cases where bleeding cannot be stopped within 5 minutes.
3. Complete pulpotomy During a total coronal pulpotomy, the coronal pulp tissue is removed down to the level of the orifices using a sterile diamond bur with copious water cooling. Bleeding is controlled by gentle pressure with a cotton pellet soaked in 2.5% NaOCl. When the bleeding stops, the cavity is flushed with sterile saline and Biodentine or MTA is applied the same way as in case of direct pulp capping. Complete pulpotomy is the treatment type of choice in the following clinical situations: (1) reversible pulpitis/normal pulp with anemic necrotic tissue in the pulp, (2) reversible pulpitis, normal pulp after partial pulpotomy if bleeding cannot be controlled in 5 minutes, (3) if the patient's complaints include spontaneous or persistent pain/night pain. Exclusion criteria for complete pulpotomy treatment include (1) bleeding uncontrollable in 5 minutes, or (2) anaemic/necrotic tissue at the level of the orifices.

The patients will be consulted about any complaints or changes in complaints 7 days after the procedure, at the same time as the final restoration is made. If there are no previous complaints, the patient will be referred back for a follow-up examination six months after the procedure. Then, after recording any complaints, a control radiograph and clinical examination (inspection, palpation, palpation, periodontal pocket probing) are performed. The same is repeated 1 year, 2 years, 3 years and 4 years after treatment. Evaluation of the results: The success of the treatment is evaluated by combining the patient's subjective complaints with the results of the clinical examination and periapical radiograph. The periapical index (PAI) is used to assess the periapical space on radiographs.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age who have at least one tooth with a pulp chamber that has been opened during a dental procedure or is likely to be opened during restoration of the tooth
* The tooth is responsive to a sensitivity test with cold spray
* The coronal part must be restorable
* The periodontal depth around the tooth should be 0 according to the Dental Practicality Index Periodontal Treatment Need, i.e. the probing depth around the tooth should not be greater than 3.5 mm

Exclusion Criteria:

* Internal/external resorption in the tooth
* If the root development of the tooth is not yet complete or if it is a deciduous tooth
* Absolute isolation cannot be performed during the procedure
* If pulp exposure does not occur even after complete removal of caries
* The crown of the tooth cannot be restored
* Periodontium surrounding tooth affected by moderate/severe marginal periodontitis (probing depth deeper than 3.5 mm)
* Pulp exposure due to traumatic injury
* Baseline radiograph shows signs of severe pulp palcification
* Periapical lesion is around the root (Periapical index of the tooth >2)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients for the study will be selected from adult patients presenting at the ambulance of the Semmelweis University Department of Restorative Dentistry and Endodontics and who meet the inclusion criteria
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
To compare the success rate between direct pulp capping, partial pulpotomy, and full pulpotomy | 4 years
  To measure the percentage of patients without any sympoms (0 on VAS scale), pain on percussion, palpation and without any radiographic sign of periapical pathosis (PAI 1 or 2)

SECONDARY OUTCOMES:
To establish a relationship between success rate, age, and other co-factors | 4 years
  The ratio of successful participants in older population, in population with systemic diseases

CONTACTS AND LOCATIONS:
Overall Officials: János Vág, DMD, PhD, Study Chair — Semmewleis University, Department of Restorative Dentistry and Endodontics
Locations (1):
- Department for Restorative Dentistry and Endodontics, Semmelweis University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elmsmari F, Ruiz XF, Miro Q, Feijoo-Pato N, Duran-Sindreu F, Olivieri JG. Outcome of Partial Pulpotomy in Cariously Exposed Posterior Permanent Teeth: A Systematic Review and Meta-analysis. J Endod. 2019 Nov;45(11):1296-1306.e3. doi: 10.1016/j.joen.2019.07.005. Epub 2019 Sep 10. PMID 31515048
- [Background] Asgary S, Eghbal MJ, Fazlyab M, Baghban AA, Ghoddusi J. Five-year results of vital pulp therapy in permanent molars with irreversible pulpitis: a non-inferiority multicenter randomized clinical trial. Clin Oral Investig. 2015 Mar;19(2):335-41. doi: 10.1007/s00784-014-1244-z. Epub 2014 Apr 27. PMID 24771228
- [Background] European Society of Endodontology (ESE) developed by:; Duncan HF, Galler KM, Tomson PL, Simon S, El-Karim I, Kundzina R, Krastl G, Dammaschke T, Fransson H, Markvart M, Zehnder M, Bjorndal L. European Society of Endodontology position statement: Management of deep caries and the exposed pulp. Int Endod J. 2019 Jul;52(7):923-934. doi: 10.1111/iej.13080. PMID 30664240